CLINICAL TRIAL: NCT02420834
Title: Dry Eye Treatment With Artificial Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DOptomEssa
Record Dates: First submitted 2015-04-10; First posted 2015-04-20 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tear Supplement Hypromellose 0.15% (Experimental): Preservative free Hypromellose Eye Drops BP 0.15% applied as required for 1 month
  Interventions: Other: Hypromellose 0.15%
- Tear Supplement Hypromellose 0.4% (Experimental): Preservative free Hypromellose Eye Drops BP 0.4% applied as required for 1 month
  Interventions: Other: Hypromellose 0.4%
- Tear Supplement Carboxymethylcellulose (Experimental): Tear Supplement 3: Preservative free 0.25% Carboxymethylcellulose, electrolyte balanced (Theratears) applied as required for 1 month
  Interventions: Other: Carboxymethylcellulose
- Tear Supplement Liposomal spray (Experimental): Preservative free Phospholipid liposomal spray (Tears Again) applied as required for 1 month
  Interventions: Other: Liposomal Spray

INTERVENTIONS:
Other: Hypromellose 0.15% — Tear supplement to be taken as required to relieve symptoms
  Other Names: Hypromellose is also sold as Isopto plain eye drops
  Arms: Tear Supplement Hypromellose 0.15%
Other: Hypromellose 0.4% — Tear supplement to be taken as required to relieve symptoms
  Other Names: Hypromellose is also sold as Isopto plain eye drops
  Arms: Tear Supplement Hypromellose 0.4%
Other: Carboxymethylcellulose — Tear supplement to be taken as required to relieve symptoms
  Other Names: Theratears
  Arms: Tear Supplement Carboxymethylcellulose
Other: Liposomal Spray — Tear supplement o be taken as required to relieve symptoms
  Other Names: Tears Again
  Arms: Tear Supplement Liposomal spray

SUMMARY:
Dry eye is a chronic irritating eye condition that affects many people, caused by poor tear quality and insufficient quantity. Treatments are traditionally in the form of artificial tears applied to the ocular surface. However, there is little evidence in the scientific literature that demonstrates their efficacy relative compared to each other, nor how to decide which one might be most effective for an individual patient. Therefore the investigators aim to examine the efficacy of different classes of artificial tears (those designed to increase viscosity, reduce evaporation or to mimic the component balance of the natural tears). In addition, the investigators also aim to determine how the treatment preferred by an individual could potentially have been predicted from their baseline condition.

DETAILED DESCRIPTION:
The efficacy of different classes of artificial tears (non-pharmaceutical) will be examined in patients that report dry eyes by prescribing each category of treatment [0.40% Sodium Hyaluronate (Clinitas Soothe), 0.15% Sodium Hyaluronate (Hyabak), 0.25% Carboxymethylcellulose, electrolyte balanced (Theratears), and Phospholipid liposomal spray (Tears Again)] for a month in turn following a short wash-out period and to examine their tear film and ocular surface after each one.

ELIGIBILITY:
Inclusion Criteria:

* subjective symptoms indicative of dry eye

Exclusion Criteria:

* Diabetes
* Sjögren's Syndrome
* recent ocular infection
* hay fever
* used any eye drops or ocular medications,
* were currently on medications known to affect the eyes
* wore contact lenses
* were pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Symptoms | 4 months
  Short questionnaire (Ocular Surface Disease Index)

SECONDARY OUTCOMES:
Non-invasive break-up time | 4 months
  Tear stability will be assessed using the Purkinje reflection from the tear film on the ocular surface recording the time (in seconds) that the reflection is first distorted, observed with a slit lamp biomicroscope
Tear meniscus height | 4 months
  Tear meniscus height will be assessed in millimetres by comparing to the slit height adjustment of a slit lamp biomicroscope.
lid parallel conjunctival folds | 4 months
  Lid parallel conjunctival folds will counted as observed with a slit lamp biomicroscope and timed/graded
Ocular Surface Staining | 4 months
  Ocular surface staining with fluorescein and lissamine green dyes will be observed with a slitlamp biomicroscope and graded using the Efron grading scale
Phenol Red Test | 4 months
  Tear volume will be quantified in millimetres after 15s with the tip inserted in the lower tear meniscus from the wetting height of a phenol red impregnated strip inserted in the lower fornix for 15 seconds

CONTACTS AND LOCATIONS:
Overall Officials: James S Wolffsohn, BSc PhD, Principal Investigator — Aston University
Locations (1):
- Specsavers, Thornton, Cleveleys, United Kingdom